CLINICAL TRIAL: NCT03316092
Title: Update on Monitoring and Preventing Hydroxychloroquine Toxicity.
Brief Title: Monitoring and Preventing Hydroxychloroquine, Plaquenil, Toxicity.
Status: Completed | Type: Observational
Sponsor: Dr. S.S. Michel Clinic (Other)
Responsible Party: Principal Investigator, Dr. Shawkat Michel, Principal Investigator, Dr. S.S. Michel Clinic
Other Study IDs: Ocular Plaquenil Toxicity
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Hydroxychloroquine Toxicity
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: optical coherence tomography — screening and monitoring all patients who are to use or have been using oral Hydroxychloroquine

SUMMARY:
Oral Hydoxychloroquine is a very popular medication widely used by patients with rheumatoid arthritis, Systemic Lupus Erythematosus and other diseases. Ocular side effects of this medication are very serious and causes loss of central vision. In most patients these side effects are dose related, cumulative. This means that the risk of side effects would increase in all patients with continued use of the medication. In few people use of the medication would not be recommended if they have some bilateral macular problems. This is because the side effects of this medication does cause serious degredation of the macula in both eyes.

DETAILED DESCRIPTION:
The ocular side effects of Hydroxychloroquine has been known for long time. Due to the seriousness of these side effects all possible efforts were done to prevent them. Preventing these side effects would ideally need prior screening of all patients who are to use oral Hydroxychloroquine. If patients are not screened prior to oral Hydroxychloroquine use they should be examined as soon as possible after starting this medication. Advances in technology, specifically the advent of optical coherence tomography, made screening and monitoring for Hydroxychloroquine toxicity much more easier and reliable meantime.

ELIGIBILITY:
Inclusion Criteria: all patients who need treatment with oral Hydroxychloroquine.

-

Exclusion Criteria: patients who are not using oral Hydroxychloroquine.

-

Ages: 25 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients whose doctors decide to treat them with oral Hydroxychloroquine. This medication is very popular in treating patients with rheumatoid arthritis and some other auto-immune diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-01-07 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
optical coherence tomography (OCT) is a very reliable, accessible and documented way for monitoring all people who are to use or have been using oral Hydroxychloroquine | Ten years
  OCT would very much help in selecting patients who may safely use oral Hydroxychloroquine. It is also the most preferred way so far for monitoring all patients who use oral Hydroxychloroquine to prevent serious and bilateral ocular side effects

CONTACTS AND LOCATIONS:
Overall Officials: shawkat s michel, FRCS Ed, Principal Investigator — Dr. S.S. Michel Clinic
Locations (1):
- Dr. S.S. Michel Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided